CLINICAL TRIAL: NCT06506877
Title: A Cognitive Risk Calculator and Screening Tool for Primary Care Settings
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Darlene Floden, Staff Neuropsychologist, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-1022; R33AG069729 (NIH)
Record Dates: First submitted 2024-07-11; First posted 2024-07-18 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Cognitive Risk Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Experimental): Active Phase: Implementation of Cognitive Risk Calculator (RC) and Brief Assessment of Cognitive Health (BACH)
  Interventions: Behavioral: Implementation of Cognitive Risk Calculator (RC) and Brief Assessment of Cognitive Health (BACH)
- Control (No Intervention): Control Phase: Prior to implementation of Cognitive Risk Calculator (RC) and Brief Assessment of Cognitive Health (BACH)

INTERVENTIONS:
Behavioral: Implementation of Cognitive Risk Calculator (RC) and Brief Assessment of Cognitive Health (BACH) — Enrolled providers will have access to two cognitive screening tools during the active phase. The first tool is a Cognitive Risk-Calculator (RC), integrated into the Electronic Health Record, to help providers identify patients who are at high risk of exhibiting cognitive decline. The second tool is a computerized cognitive screening tool, the Brief Assessment of Cognitive Health (BACH), which patients complete independently. Results are automatically entered into the patient's medical record, along with patient-specific flags for concerns about depression and/or sleep disorder. The purpose of these tools is to facilitate cognitive screening and treatment for factors that may be contributing to cognitive decline.
  Arms: Active

SUMMARY:
This mixed-methods pragmatic trial will use a stepped wedge cluster randomized design to implement a cognitive risk-calculator and automated cognitive screening tool (BACH) in eight internal medicine clinics in the Cleveland Clinic Health System. Administrative and EHR data will provide quantitative metrics of adoption (tool use) and effectiveness (change in provider behavior) while observations, interviews, and questionnaires will assess fidelity, acceptability, and feasibility for all stakeholders. Analyses will consider provider characteristics, clinic attributes, and regional variations in patient characteristics (e.g., SES, race/ethnicity).

ELIGIBILITY:
Provider Inclusion Criteria:

* Must see adults aged 60 years or older in their practice.
* Must be a prescribing provider.

Exclusion Criteria:

* Provider sees patients at more than one participating study site.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Adoption of RC and BACH: Frequency of Cognitive Screening | Monthly assessment over the study duration (up to 1 year)
  Number of cognitive screening events per month, stratified by screening tool (BACH vs other) and Risk Calculator category (high vs low risk).
Adoption of RC and BACH: Frequency of BACH Orders | Monthly assessment over the study duration (up to 1 year)
  Number of BACH orders or pre-visit order sets executed per month, stratified by Risk Calculator category (high vs low risk).
Effectiveness of RC and BACH: Frequency of MCI/ADRD, Sleep Disorders, and Depression Diagnoses | Monthly assessment over the study duration (up to 1 year)
  Incidence of new diagnoses for cognitive impairment (including MCI and ADRD), sleep disorders, and depression per month, stratified by screening completed (BACH/other/none) and Risk Calculator category (high vs low risk).
Effectiveness of RC and BACH: Frequency of Referrals to Neuropsychology, Geriatrics/Neurology, Psychiatry/Psychology, and Sleep Medicine | Monthly assessment over the study duration (up to 1 year)
  Number of orders and consults placed to specialty services per month, stratified by screening completed (BACH/other/none) and Risk Calculator category (high vs low risk).
Effectiveness of RC and BACH: Prescription Rates for Related Medications | Monthly assessment over the study duration (up to 1 year)
  Number of new medication orders relevant to cognition, sleep, and mood per month, stratified by screening completed (BACH/other/none) and Risk Calculator category (high vs low risk).

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No